CLINICAL TRIAL: NCT06093256
Title: Orthodontic Fixed Appliances' Impact on Taste Perception Among Orthodontic Patients: A Prospective Cohort Study
Brief Title: Taste Changes With Fixed Orthodontic Appliances
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Hassan Geza A AlHarby, Postgraduate student, Riyadh Elm University
Other Study IDs: Taste changes and ortho
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Taste Perception; Fixed Orthodontic Appliances
Keywords: Fixed Orthodontic Appliances; Taste Alterations; Taste Perception
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fixed orthodontic appliances — Taste sensation will be checked before and after fixed orthodontic therapy.

SUMMARY:
The aim of this research:

1. To analyze the possible influence of fixed orthodontic appliances on taste perception among patients undergoing conventional orthodontic treatment.
2. To objectively assess taste perception in patients with fixed orthodontic appliances using taste strips.

DETAILED DESCRIPTION:
Orthodontic treatment has become the most common therapy among dental treatment seekers, with wide-ranging implications for oral health and overall quality of life. Malocclusion, if left untreated, can lead to various functional and aesthetic issues, including chewing difficulty, speech problems, increased risk of caries, and compromised facial aesthetics, which can significantly impact an individual's quality of life. In addition, the aesthetic impact of malocclusion can affect individuals' self-esteem, social interactions, and psychological well-being. So, malocclusion and correction of the same have become a priority. The prevalence of malocclusion varies among different populations and geographical regions. Factors such as genetics, ethnicity, and environmental influences contribute to these variations. In Saudi Arabia, malocclusion prevalence is significantly high, with crowding of teeth being the most common type, followed by teeth spacing, along with excessive overjet and overbite. Conventional fixed orthodontic treatment, involving brackets and wires, is a widely accepted approach to correct malocclusions. This treatment modality aims to move the teeth into proper alignment, correct bite discrepancies, and achieve optimal occlusion. Moreover, it has long been recognized as a highly effective treatment approach for correcting malocclusion.

In orthodontic therapy, much attention is devoted to the alignment and aesthetics of teeth. However, one aspect that often goes overlooked is the potential alteration of taste perception. According to Bernabé (2008), orthodontically treated patients with fixed appliances reported food intake difficulties. In addition, placing these appliances in the mouth may interfere with or alter the sense of taste. Proper perception of taste, as one of the most important sensual sensations, contributes significantly to human well-being, both in the physical and mental senses, which is a health condition as defined by the WHO. Impaired perception of taste stimuli may occur as a result of a foreign body placement such as placement of the orthodontic material in the oral cavity. Therefore, from a clinical point of view, evaluating the relationship between using fixed orthodontic appliances and its impact on the sense of taste is of greater importance. Taste perception or gustation is a multisensory experience that helps in the sensory recognition of food on the tongue and plays a fundamental role in determining the flavors of foods. In humans, the sensation of taste can be categorized as salty, sour, bitter, sweet, and umami. Alteration or loss of gustation may arise due to a wide range of systemic or acute clinical conditions or medications. Therefore, testing this alteration or loss of taste sensation has become a common mode. One of the simple assessments of taste senses is by using the taste strips as described by Mueller and colleagues. These strips are composed of filter paper and soaked with different taste solutions. A review of the literature to date on taste perception has yielded only a few reports. Further, no reports have been published regarding the altered taste perception and flavor after fixed orthodontic treatment. Thus, this study aims to evaluate changes in taste perception after conventional fixed orthodontic appliance treatment. The outcome of this investigation on the alterations in taste perception and exploring the potential mechanisms will deepen our understanding of the comprehensive effects of orthodontic treatment and enhance patient satisfaction and quality of life.

Most studies in the literature have evaluated the changes in taste sensation using removable orthodontic appliances. Yet, studies on conventional fixed appliances are insufficient. Two studies analyzed taste alterations using removable orthodontic appliances, showing no significant difference in taste perception between patients with and without orthodontic appliances. These findings could be attributed to their short duration of wear, ease of removal, and the fact that appliances could be kept outside the mouth during meals. Wilczyska et al. (2011) conducted the sole study investigating palatal fixed auxiliary appliances' impact on taste perception. They have reported that the identification and perception of different taste sensations and the duration of a taste stimuli reaction were not affected by these appliances. Hence, there was no evidence that the studied orthodontic devices had impaired taste abilities. Another study by Razdan et al. (2017) has shown that there was a transient change in taste perception during the use of removable orthodontic appliances, but this change did not significantly affect taste stimuli.

Nevertheless, there was one study that examined the discomfort experienced by patients with conventional fixed orthodontic appliances, and the results of the study indicated a significant relationship between orthodontic fixed appliances and taste impairment. Overall, it is clear from the review that there is a conflicting report on the effect of orthodontic appliances on the perception of taste. Therefore, the present study is aimed at assessing changes in taste perception after conventional fixed orthodontic appliance treatment.

This proposal aims to shed light on this intriguing phenomenon and its implications for orthodontic care. By investigating the alterations in taste perception and exploring potential mechanisms behind these changes, we can deepen our understanding of the comprehensive effects of orthodontic treatment and enhance patient satisfaction and quality of life.

Material and Methods:

Research design This is an in-vivo clinical study (prospective cohort) that will be conducted at Ortho-Pedo Centre (Riyadh Elm University) to analyze the gustatory perception and alteration in patients undergoing fixed orthodontic treatment. Both genders with ages ranging from 15 to 35 years old will be included in this study. Authorizing their participation by signing the informed consent.

Method of assessment A self-administered questionnaire will be used before and after the orthodontic treatment to assess taste perception.

The material used to assess the alteration in the taste function:

To assess the taste function, the paper filter strips ("Taste Strips", Burghart, Wedel, Germany) will be used. This strip clinically assesses the taste's function by using four concentrations with a maximum total score of 16 and 4 for each taste quality, resulting in a maximum total score of 16 and 4 for each taste quality.

Method of using the strips The taste strips (plus two blank strips devoid of flavor) will be applied on the extending tongue immediately posterior to its first third, either to the left or right, for the purpose of examining lateralization. In order to proceed, participants will be required to seal their lips and select one of five possibilities (sweet, sour, salty, bitter, or no taste). To distinguish different taste perceptions, they will be instructed to rinse their mouths with water before evaluating each flavor strip.

The method of assessment: the course of examination

* It will be ensured that all the subjects will avoid eating or drinking anything other than water two hours before testing.
* Patients will also be advised not to smoke and not to brush their teeth.
* The 16 taste strips are presented to the patient in a 'pseudo-randomized' order, one after the other. The patient will be instructed to rinse their mouth thoroughly with clean water in between strips. The exam will be administered alternately to the left and right sides, on each side independently.
* The patient will be requested to select one response from the following options: 1. sweet, 2. salty, 3. bitter, 4. sour, and 5. no taste.
* Each correct answer will be given one point. Thus, the maximum score is 4 for each taste quality or 16 for the definite test.
* Along with the impregnated strips, two strips with no taste (blanks U + V) can be integrated into the examination at any time (no points).

Labeling of the Taste Strips and containers:

The Taste Strips and the containers are consecutively numbered from A - P and U + V as shown in this figure:

Normal values received from young, healthy test persons for the complete mouth test range from 9-16 points.

The time period for the assessment of taste

* T0 - 2 weeks prior to bonding of the fixed appliance (baseline).
* T1 - Immediately after bonding of the fixed appliance.
* T2 - 13 weeks after appliance installation. All clinical measurements will be conducted by one single examiner.

Statistical analysis Data obtained will be analyzed using the SPSS (Version 20.0, Chicago, Illinois) software. The descriptive data will be expressed in terms of means with standard deviations and percentages. Shapiro Wilk test of normality will be used to determine the distribution of the continuous data. A parametric (ANOVA) test will be used if the data is normally distributed and a non-parametric (Kruskal Wallis) test will be used if the data is skewed. Chi-square and Fisher Exact tests will be employed to assess the association between the variables. Statistical significance will be set at p ≤ .05.

Ethical approval The study will be submitted to the institutional review board (IRB) at Riyadh Elm University (REU) and will follow REU's IRB policies and procedures.

Verbal consent will be obtained from the participants before data collection and using the Burghart taste strips. Detailed information will be provided about the aim and benefits of the study. All patients will be informed that their participation is voluntary. Anonymity and confidentiality will be ensured.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in orthodontic therapy by conventional fixed orthodontic treatment.
2. At least aged 15 years and over.

Exclusion Criteria:

1. Any patients with endocrine abnormalities (diabetes mellitus, thyroid gland dysfunction, Cushing's disease).
2. Any internal disorders (chronic renal failure, liver cirrhosis)
3. Middle ear infections.
4. Smoking patients.
5. Depression and xerostomia.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total sample of 40 volunteers will be studied at 3 different time points. The sample size for the study was calculated based on the medium effect size obtained from the study by Mueller et al. (2003) by considering α error probability (0.05) and required power (1-β err prob) (0.93). While keeping in mind the resources and time limits to conduct the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of taste perception with the use of fixed orthodontic appliances | Baseline and after 13 weeks
  Analysis of taste changes before and after orthodontic treatment using taste filter strips.

REFERENCES:
- [Background] Ajwa N, AlHammad A, AlAmmar L, AlMarjan M, AlShugair T, AlManie L, Bangalore D. The Influence of Orthodontic Treatment Need on Oral Health-Related Quality of Life among 12-18-Year-Old Adolescents in Riyadh. Healthcare (Basel). 2022 Oct 28;10(11):2153. doi: 10.3390/healthcare10112153. PMID 36360492
- [Background] Almotairy N, Almutairi F. A Nation-wide Prevalence of Malocclusion Traits in Saudi Arabia: A Systematic Review. J Int Soc Prev Community Dent. 2022 Jan 29;12(1):1-11. doi: 10.4103/jispcd.JISPCD_251_21. eCollection 2022 Jan-Feb. PMID 35281679
- [Background] Bernabe E, Sheiham A, de Oliveira CM. Impacts on daily performances related to wearing orthodontic appliances. Angle Orthod. 2008 May;78(3):482-6. doi: 10.2319/050207-212.1. PMID 18416624
- [Background] Cenzato N, Nobili A, Maspero C. Prevalence of Dental Malocclusions in Different Geographical Areas: Scoping Review. Dent J (Basel). 2021 Oct 11;9(10):117. doi: 10.3390/dj9100117. PMID 34677179
- [Background] Devanna R, Felemban NH, Althomali Y, Battepati PM, Ali Alfawzan A, Gupta P. Prevalence of malocclusion among children of the Kingdom of Saudi Arabia - A systematic review and meta-analysis. Saudi Dent J. 2021 Dec;33(8):826-834. doi: 10.1016/j.sdentj.2021.09.005. Epub 2021 Sep 14. PMID 34938022
- [Background] Grewal H, Sapawat P, Modi P, Aggarwal S. Psychological impact of orthodontic treatment on quality of life - A longitudinal study. Int Orthod. 2019 Jun;17(2):269-276. doi: 10.1016/j.ortho.2019.03.009. Epub 2019 Apr 23. PMID 31028017
- [Background] Har-Zion G, Brin I, Steiner J. Psychophysical testing of taste and flavour reactivity in young patients undergoing treatment with removable orthodontic appliances. Eur J Orthod. 2004 Feb;26(1):73-8. doi: 10.1093/ejo/26.1.73. PMID 14994885
- [Background] Hassan AH, Amin Hel-S. Association of orthodontic treatment needs and oral health-related quality of life in young adults. Am J Orthod Dentofacial Orthop. 2010 Jan;137(1):42-7. doi: 10.1016/j.ajodo.2008.02.024. PMID 20122429
- [Background] Hegde AM, Dwivedi S. Effect of removable orthodontic appliance on taste and flavor perception--a clinical study. J Clin Pediatr Dent. 2007 Fall;32(1):79-82. doi: 10.17796/jcpd.32.1.jt1677554845122u. PMID 18274477
- [Background] Izabella Dunin-Wilczyńska1, ,. U. Ż. A. M. T. B., (2011). Effects of Palatal Fixed Auxiliary Appliances on the Sense of Taste. Dental and Medical Problems, Volume 48, p. 217-222. https://dmp.umw.edu.pl/en/article/2011/48/2/217/
- [Background] Kiyak HA. Does orthodontic treatment affect patients' quality of life? J Dent Educ. 2008 Aug;72(8):886-94. PMID 18676797
- [Background] Mueller C, Kallert S, Renner B, Stiassny K, Temmel AF, Hummel T, Kobal G. Quantitative assessment of gustatory function in a clinical context using impregnated "taste strips". Rhinology. 2003 Mar;41(1):2-6. PMID 12677732
- [Background] Marques LS, Paiva SM, Vieira-Andrade RG, Pereira LJ, Ramos-Jorge ML. Discomfort associated with fixed orthodontic appliances: determinant factors and influence on quality of life. Dental Press J Orthod. 2014 May-Jun;19(3):102-7. doi: 10.1590/2176-9451.19.3.102-107.oar. PMID 25162573
- [Background] Proffit, W. R., Fields, H. W., Larson, B. E., & Sarver, D. M. (2019). Contemporary Orthodontics. Philadelphia, PA: Elsevier. https://shop.elsevier.com/books/contemporary-orthodontics/proffit/978-0-323-54387-3
- [Background] Razdan P, Sakthivel VS, Naqvi ZA, Goyal V, Tripathi S, Singh S. Alteration in Taste Perception among Young Children during the use of Removable Orthodontic Appliance Therapy. J Contemp Dent Pract. 2017 Jul 1;18(7):607-613. doi: 10.5005/jp-journals-10024-2093. PMID 28713117
- [Background] Sergl HG, Zentner A. A comparative assessment of acceptance of different types of functional appliances. Eur J Orthod. 1998 Oct;20(5):517-24. doi: 10.1093/ejo/20.5.517. PMID 9825554
- [Background] Spence C. Multisensory flavor perception. Cell. 2015 Mar 26;161(1):24-35. doi: 10.1016/j.cell.2015.03.007. PMID 25815982
- [Background] Stewart FN, Kerr WJ, Taylor PJ. Appliance wear: the patient's point of view. Eur J Orthod. 1997 Aug;19(4):377-82. doi: 10.1093/ejo/19.4.377. PMID 9308258
- [Background] Taruno A, Nomura K, Kusakizako T, Ma Z, Nureki O, Foskett JK. Taste transduction and channel synapses in taste buds. Pflugers Arch. 2021 Jan;473(1):3-13. doi: 10.1007/s00424-020-02464-4. Epub 2020 Sep 16. PMID 32936320